CLINICAL TRIAL: NCT06669507
Title: The Sleep Clinic Outcome and Practice Study: The SUP-study
Brief Title: The Sleep Clinic Outcome and Practice Study
Acronym: SUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 710756
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Insomnia Disorder; Circadian Rhythm Sleep Disorder
Keywords: Insomnia Disorder; Circadian Rhythm Sleep Disorder; Sleep treatment; CBT-I; Chronotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm | interventions — Chronotherapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Non-randomized single-arm treatment study with treatment as usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment as usual (Other): All patients referred to the Sleep Clinic and that is considered eligible and has a signed consent will be included in the study.
  Interventions: Behavioral: Chronotherapy; Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Chronotherapy — 1. The effect of light exposure follows a phase-response curve where circadian phase advancement is strongest in the biological morning, whereas light in the biological evening/night may lead to a phase delay. Light therapy is provided by 30 min light exposure using 10 000 lux light boxes.
  2. Melatonin 3 milligram is prescribed in tablet forms (not depot), usually 12 hours before the planned rise time.
  3. Additionally, blue-light-blocking glasses are used to block light exposure at night, which has been found to advance circadian rhythms. Patients are advised to wear their blue-blocking glasses 12 hours before rise time.
  Which chronotherapeutic interventions that are used, is considered individually by the clinicians in the Sleep Clinic, but often all three treatment components are used at the same time. Duration of chronotherapy given in the Sleep Clinic vary from 4 to 8 consultations over 1 to 4 months depending on the patients' needs and progress during treatment.
Behavioral: Cognitive Behavioral Therapy for Insomnia — All participants will receive treatment as usual. CBT-I has several components and consists of the following interventions including psychoeducation about sleep: sleep hygiene, sleep restriction therapy, stimulus control, and challenging beliefs and perceptions of sleep. Special emphasis is placed on providing a rationale for behavior change as a primary means of improving sleep as well as addressing dysfunctional beliefs the patients may hold about sleep. During treatment, tapering sleep medication is not necessary. However, if the patients are motivated to do so, this is discussed and a plan for tapering is provided. Treatment duration is typically between 4 to 8 consultations over 1 to 4 months depending on the patients' needs and progress during treatment.
  Other Names: CBT-I

SUMMARY:
The goal of this clinical trial is to explore the outcome and practice treatment for sleep-wake disturbances in a Sleep Clinic. The main questions it aims to answer are:

* What is the practice (timing and duration of treatment components) of sleep-wake disturbance treatment?
* What is the treatment effect of sleep-wake disturbance treatment.

Participants will receive treatment as usual by consultations with a trained psychiatrist or psychologist and will be asked to fill out self-reporting questionnaires and sleep diaries.

DETAILED DESCRIPTION:
Background: Sleep-wake disturbances including insomnia disorder and sleep-wake rhythm disorders disables many aspects of life and is highly prevalent. As one of few treatment options for sleep-wake disturbances, the Sleep Clinic at St. Olavs Hospital offers clinical assessments and treatment for this patient group in Norway. Although the treatment of insomnia disorder is well-described and recommended, there is still a major subgroup that to not benefit from the treatment. Additionally, treatment and outcome of sleep-wake rhythm disorders is little described in clinical settings. A study of clinical practice and outcomes of the treatments in the Sleep Clinic, would give the possibility to illuminate these knowledge gaps.

Aim: Describe the practice (timing and duration) and outcomes of the sleep treatments 1) Cognitive Behavioral Therapy for Insomnia and 2) Chronotherapy for sleep-wake rhythm disorders at the Sleep Clinic at St. Olavs Hospital.

Method: All patients referred to the Sleep Clinic will be asked to participate before the first consultation with a clinician. Patients will be clinically assessed, diagnosed and given treatment as usual. Main outcomes will be self-report questionnaires at treatment termination and the use, timing and duration of specific sleep treatment components logged by the clinician during treatment.

Potential impact: The findings from this research project provides possibilities to improve treatment for sleep-wake disturbances by tailoring the treatment different to respective subgroups. The findings will also contribute to novel knowledge on how to treat patients with sleep-wake rhythm disorders and to what degree they benefit from the treatment in a sleep clinic.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the Sleep Clinic at St. Olavs Hospital for an assessment of a sleep-wake disruption.
* Age >= 18 years.
* Willing and able to provide written informed consent.
* Meeting the diagnostic criteria for at least one of the following disorders: F51.0 Insomnia disorder or G47.2 Sleep-wake rhythm disorders, considered being either: Delayed sleep-wake phase disorder, Advanced sleep-wake phase disorder, Non-24-hour sleep-wake disorder or Irregular sleep-wake disorder
* Desire non-pharmacological sleep treatment

Exclusion Criteria:

* Individuals working night shifts or that otherwise have external conditions that result in inadequate sleep opportunity, such as caring for an infant or does not have permanent housing etc.
* Individuals being blind
* Individuals being psychotic
* Individuals having epilepsy
* Individuals having an ongoing substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep treatment practice | Through study completion, an average of 8 weeks.
  Timing and duration of sleep treatment componements
Sleep treatment outcome | Through study completion, an average of 8 weeks.
  1. Insomnia Severity Index for insomnia disorder
  2. Insomnia Severity Index with additional question for sleep-wake rhythm disorders

SECONDARY OUTCOMES:
Testing the effectiveness of sleep treatment outcomes in different modes of treatment delivery | Through study completion, an average of 8 weeks.
  1. Group versus individual delivery of sleep treatment.
  2. Telemedicine versus face-to-face delivery of sleep treatment

CONTACTS AND LOCATIONS:
Overall Officials: Knut Langsrud, PhD/MD, Study Director — St. Olavs Hospital
Locations (1):
- Sleep Clinic, St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD outside the research team in Trondheim.

DOCUMENTS (2):
  • Study Protocol (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT06669507/Prot_000.pdf
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT06669507/ICF_001.pdf